CLINICAL TRIAL: NCT00000587
Title: Erythropoietin for Anemia Due to Zidovudine in Human Immunodeficiency Virus Infection
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Thomas Jefferson University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Masking: Double | Purpose: Treatment
Other Study IDs: 307
Record Dates: First submitted 1999-10-27; First posted 1999-10-28 (Estimated); Last update posted 2021-11-26 (Actual); Status verified 2021-11

CONDITIONS: Acquired Immunodeficiency Syndrome; Anemia; Hematologic Diseases; HIV Infections; Blood Disease
MeSH Terms: conditions — Acquired Immunodeficiency Syndrome; Anemia; Hematologic Diseases; HIV Infections | interventions — Erythropoietin

INTERVENTIONS:
Procedure: erythropoietin, recombinant

SUMMARY:
To determine whether administration of human recombinant erythropoietin (REPO) improved or eliminated the anemia seen in human immunodeficiency virus (HIV) infected patients after therapy with zidovudine (ZDV).

DETAILED DESCRIPTION:
BACKGROUND:

Reports had shown that between 24 and 78 percent of patients with Acquired Immune Deficiency Syndrome treated with zidovudine for four to six months developed significant bone marrow toxicity, requiring zidovudine dosage alterations, blood transfusions, or cessation of therapy. While zidovudine efficacy had been demonstrated in patients with AIDS or ARC, it was also evaluated in patients with AIDS-related illness, as well as in asymptomatic HIV-infected individuals. The clinically significant zidovudine-induced anemia developing in a substantial number of these patient groups and requiring blood transfusions could cause a significant drain on the blood supply in the United States.

The project was part of an Institute-initiated study on the Pathobiology of Bone Marrow Suppression in AIDS or AIDS-Related Complex. The concept was approved at the May 1987 National Heart, Lung, and Blood Advisory Council. The Request for Applications was released in December 1987.

DESIGN NARRATIVE:

Double-blind, placebo-controlled. Patients received intravenous REPO (1000 IU/kg) or placebo twice per week. The five patients in Group A had no transfusion history. The five patients in Group B had a history of transfusions. Prior to the study, the authors determined that treatment would continue for twelve weeks or until the hemoglobin reached 12.5 g/dl. After the twelve week study period, patients were eligible to receive open label erythropoietin (500 IU/kg, twice a week). For numerous reasons, recruitment of patients was a major problem in this trial. The study originally estimated a total of 64 patients.

ELIGIBILITY:
No eligibility criteria

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Dates: Start 1988-09 (Actual); Primary Completion 2005-01 (Actual); Study Completion 2005-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Stephen Hauptman — Jefferson Medical College of Thomas Jefferson University